CLINICAL TRIAL: NCT05192018
Title: Reversal of a Defunctioning Ileostomy 3 Weeks After the Index Operation, RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Debakey3
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): This group will have their ileostomy reversed after 3 weeks from the index operation. All procedures were performed by the same senior surgeons. The duration of the operation was noted and the ease of reversal of stoma and closure of abdominal wall were assessed on ascale of 0-10 (0 = difficult, 10 = easy) by the operating surgeons.
  Interventions: Procedure: Early reversal of a defunctiong ileostomy
- Group B (Active Comparator): This group will be discharged home after the primary colorectal surgery with a defunctioning ileostomy and brought back after an interval of 3 months ,or after completion of their adjuvant therapy, for reversal. All procedures were performed by the same senior surgeons. The duration of the operation was noted and the ease of reversal of stoma and closure of abdominal wall were assessed on ascale of 0-10 (0 = difficult, 10 = easy) by the operating surgeons.
  Interventions: Procedure: Early reversal of a defunctiong ileostomy

INTERVENTIONS:
Procedure: Early reversal of a defunctiong ileostomy — Early reversal of a defunctiong ileostomy after 3 weeks of its creation

SUMMARY:
Diverting ileostomy seems to mitigate the consequences of anastomotic leak from low rectal anastomosis. Gastrointestinal continuity is restored after a period of 6-12 weeks but it can be longer if the patient is on adjuvant chemotherapy or due to low priority given to this procedure. This exposes up to one-third of the patients to significant morbidity having an impact on the quality of life and considerable economic costs. Although no meta-analysis data determined the safety and optimal time for the closure of a temporary diversion of the small bowel, earlier reversal of ileostomies a few days after primary anastomosis reduces the length of exposure to stoma-related morbidity and may improve quality of life, reduce stoma-related costs and still protect the distal anastomosis. Herein, we aimed to assess the results of early closure of defunctioning ileostomy a week following a satisfactory anastomosis, negative air leak test and smooth post-operative course and in absence of worrisome clinical signs of anastomotic leak with optional intraoperative visualization of the anastomostic line by endoscopy immediately before closing the ileostomy.

DETAILED DESCRIPTION:
All consecutive patients coming to National Cancer Institute of Cairo university, having a defunctioning ileostomy during a low rectal or anal anastomosis or even for obstructive purposes, will be considered eligible and offered to participate in the trial. Patients currently on steroids, at high cardiorespiratory risk and those experiencing any postoperative complication will be excluded. Informed written consent will be obtained from the patients. The remaining patients were randomized into early (Group A) and late (Group B) reversal groups using sealed envelopes. Group A will have their ileostomy reversed after 3 weeks from the index operation within one hospital admission, while group B will be discharged home and brought back after an interval of 3 months ,or after completion of their adjuvant therapy, for reversal. All procedures were performed by the same senior surgeons. The duration of the operation was noted and the ease of reversal of stoma and closure of abdominal wall were assessed on ascale of 0-10 (0 = difficult, 10 = easy) by the operating surgeons. Postoperative complications were recorded in concordance with the definitions of Dindo et al. [5]. Costs associated with stoma care (consumables and nurse visits)were calculated. Baseline and preoperative characteristics of the patients. Baseline demographics (age, gender, ECOG score, smoking, DM, BMI) and immediate postoperative outcome (complications, if any, like anastomotic leakage, ileus, wound problems and others, rate of reoperation, and 30-day mortality) will be analyzed as well.

Exclusion criteria

* When performed to cover unsatisfactory anastomosis
* Positive air-leak test
* Those experienced postoperative complications
* Those with preoperative (1st operation) albumin below 3.5gm/dL.
* Immunocompromised patients e.g on steroids or have uncontrolled DM.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have a defunctioning ileostomy after a colorectal surgery

Exclusion Criteria:

* When performed to cover unsatisfactory anastomosis
* Positive air-leak test
* Those experienced postoperative complications
* Those with preoperative (1st operation) albumin below 3.5gm/dL.
* Immunocompromised patients e.g on steroids or have uncontrolled DM.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-25 (Actual); Primary Completion 2023-07-25 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
Feasibility of early reversal of adefunctioning ileostomy | 1 month after the operation
  Feasibility will be measured by recording post operative complications according to Clavien- Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mahmoud, Professor, Study Director — National Cancer Institute, Cairo University, Egypt
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
In a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication and for a year
Access Criteria: In the Journal of publication